CLINICAL TRIAL: NCT05797090
Title: Comparative Study Between Conventional Crystalloid Cardioplegic Solution With Modified Del Nido Cardioplegia in Mitral Valve Regurgitation Surgery
Brief Title: Comparative Study Between Conventional Crystalloid Cardioplegic Solution With Modified Del Nido Cardioplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mohamed (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor-Investigator, mohamed, Lecturer of Anesthesia, intensive care and pain management Faculty of Medicine - Al-Azhar University, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Moustafa Omara
Record Dates: First submitted 2023-02-25; First posted 2023-04-04 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Mitral Valve Surgery
MeSH Terms: interventions — potassium cardioplegic solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- crystalloid cardioplegia with modified del Nido cardioplegia (Experimental): To compare between conventional crystalloid cardioplegia with modified del Nido cardioplegia in mitral valve regurge replacement surgery.
  Interventions: Drug: Crystalloid Cardioplegic solution

INTERVENTIONS:
Drug: Crystalloid Cardioplegic solution — To compare between conventional crystalloid cardioplegia with modified del Nido cardioplegia in mitral valve regurge replacement surgery.
  Other Names: Modified Del Nido Cardioplegia

SUMMARY:
Mitral valvuloplasty for correction of chronic mitral regurgitation carries a lower operative mortality and morbidity and improved long-term survival than does mitral valve replacement. Unfortunately, mitral valvuloplasty is not possible in all patients with chronic mitral regurgitation because of unfavorable pathology or lack of experience with this technique

DETAILED DESCRIPTION:
Cardioplegia is a fundamental component in providing heart protection, limiting metabolic activity and increasing the myocardium's capacity to resist ischemia for prolonged periods, thus being essential for good surgical outcomes.

Numerous cardioplegia solutions exist with different compositions to provide sufficient myocardial protection. However, there is no standard for the optimal or ideal composition and delivery technique. Cardioplegia solutions are crystalloid or blood-based solutions with various chemical compounds.

Despite improvements in myocardial protection, prosthetic valves, surgical techniques, and postoperative care, the operative mortality and morbidity of mitral valve replacement for chronic mitral regurgitation remains high in comparison with other commonly performed heart operations.

The timing of the administration of cardioplegia is extremely important in terms of preventing myocardial dysfunction. Conventional multidose cardioplegias should be repeatedly administered in every 15 to 20 min. Frequent interruption of the surgical process, even for a short time, before each cardioplegia delivery leads to a loss of time during open heart surgery, where time is extremely important, and disrupts the coherence of the operation and the surgical concentration.

Crystalloid cardioplegic solutions achieve cardioplegic arrest through inhibition of either fast-acting sodium channels or calcium-activated mechanisms. Hyperkalemia can be used to inhibit the fast-acting sodium channels as it is in the St.Thomas Hospital solution and its modifications.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for elective Mitral regurge replacement Surgery with normal Coronaries

Exclusion Criteria:

1. Patients with chronic renal disease (previous medical diagnosis or serum creatinine greater than 1.5mg/dL)
2. Left ventricular ejection fraction less than 50%.
3. Previous cardiac surgery
4. Patient with BMI > 30
5. Severe psychiatric illness
6. Inability or unwillingness to give informed consent for participation

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
myocardial protection | from baseline to 24 hours after the operation
  Number of Participants With myocardial protection through measurements of the serum levels of the cardiac enzymes just after operation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel-Gawad, Lecturer, Principal Investigator — Faculty of Medicine - Al-Azhar University
Locations (1):
- Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided